CLINICAL TRIAL: NCT05635929
Title: Effect of a Novel Topical Composition on the Incidence of Severe Oral Mucositis in Head & Neck Cancer Radiated Patients and Quality of Life Assessed by PROMs. A Two Phases Study, Part of STOP OM PROJECT. Phase 2, Single Arm, Interventional, Longitudinal, Clinical Trial.
Brief Title: Effect of a Novel Topical Composition on the Incidence of Severe Oral Mucositis in Head & Neck Cancer Radiated Patients and Quality of Life Assessed by PROMs.
Acronym: STOPOMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mucosa Innovations, S.L. (Industry)
Collaborators: HM Sanchinarro University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STOPOM01
Record Dates: First submitted 2022-11-08; First posted 2022-12-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Oral Mucositis; Quality of Life; Mucositis; Pain; Speech; Saliva; Radiation Toxicity; Chemotherapeutic Toxicity; Head and Neck Cancer
Keywords: Oral Mucositis; Cancer Therapy Toxic Effect; Cancer Support; Pain; Ulcers; Treatment Interruptions; Oral Mucosa; Radiotherapy; Chemotherapy; Head and Neck Cancer; Severe Oral Mucositis
MeSH Terms: conditions — Stomatitis; Mucositis; Pain; Speech; Radiation Injuries; Head and Neck Neoplasms; Ulcer | interventions — Betaine; Xylitol

STUDY DESIGN:
Intervention Model Description: Single group, interventional, open-label study.
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acute and Chronic outcomes in radiotherapy treated HNC patients using XCM-OM118. (Experimental): Incidence and time to onset of severe oral mucositis during radiotherapy for HNC (Acute-phase 1).
  Oral Mucositis in Head and Neck cancer patients using XCM-OM118 during radiotherapy was assessed by the clinician once weekly using the WHO scale and severity, if any, was graded from 0 to 4. Incidence and time to onset of severe oral mucositis were determined. Patient reported outcomes regarding their oral mucositis experience (pain and functional impairment) were collected through a questionnaire.
  QoL in HNC was assessed 6 months after radiotherapy and 1 month of use of XCM-OM118 (Chronic-phase 2).
  Patients who had completed oncological treatment six months earlier used the XCM-OM118 composition for one month. Quality of life was assessed at baseline and after the intervention using the University of Washington Quality of Life (UW-QOL) PROMs questionnaire, which measures domains including pain, appearance, and personal activity. Baseline scores were compared with final PROMs scores.
  Interventions: Other: XCM-OM118 Composition comprising olive oil, betaine and xylitol

INTERVENTIONS:
Other: XCM-OM118 Composition comprising olive oil, betaine and xylitol — Topical composition in the form of a gel and a mouthwash.

SUMMARY:
The use of a novel topical mucosa composition (XCM-OM118) comprising 2-(trimethylazaniumyl) acetate; (2R,3R,4S)-pentane-1,2,3,4,5-pentol; Hexadecanoic acid; (9Z, 12Z)-octadeca-9,12-dienoic acid; octadecanoic acid; (Z)-hexadec-9-enoic acid; (Z)-octadec-9-enoic acid) delivered as a gel and a mouthwash is to be studied in regard to its effect on the incidence of severe oral mucositis in Head & Neck cancer radiated patients. Patient reported outcome measures seem to be an effective tool to obtain a greater knowledge of the physical and emotional state of patients, being used in this study to assess quality of life of Head & Neck cancer radiated patients.

DETAILED DESCRIPTION:
This study analyses the severity of oral mucositis in H&N cancer patients along the first 6 weeks of radiotherapy with or without chemotherapy (Phase 1).

Phase 2 evaluates Quality of Life in a pool in H&N cancer patients 6 months after cancer treatment is completed. Quality of life of patients is analyzed before (baseline) and after 1 month period of use of the tested composition beginning 6 months after oncological treatment completion.

During cancer treatment (Phase 1), mucositis may affect the course of therapy and long-term survival, while after treatment (Phase 2) chronic pain, xerostomia, dysphagia and speech limitations between others are behind anxiety and poor quality of life.

The WHO oral mucositis scale together with a structured qualitative questionnaire to recover patient reported symptoms are used during phase 1.

A validated Quality of Life PROMS questionnaire described by the University of Washington, is chosen for Phase 2 evaluation.

Oral mucosa management is homogenized both during acute and chronic phase with the use of a novel composition comprising XCM-OM118 delivered in the form of a topical non-rinsing gel and a mouthwash.

During Phase 1, patients apply two pumps of the gel before bedtime, mid-morning, and mid-afternoon, as well as before and after each therapy session.

Six months after oncological treatment (Phase 2), patients will complete a questionnaire to assess their quality of life before implementing the oral care protocol (baseline). After 1-month intervention, patients will complete a final questionnaire.

This intervention will consist of applying two pumps of the gel before bedtime, mid-morning, and mid-afternoon. Patients will rinse with the mouthwash three times a day, ideally after brushing.

Adverse effects, such as allergic reaction, skin and/or mucosa irritation, itching, discomfort, yeast infection, or any other, will be collected and if so, a detailed description and follow-up of the problem will be noted.

ELIGIBILITY:
Inclusion Criteria:

Acute Phase

* Patients diagnosed with Head & Neck cancer who will undergo radiotherapy (with or without concomitant chemotherapy)
* Patients who are able to read, understand, and complete the questionnaire.
* Patients over 18 years of age.

Chronic Phase

* Patients who have completed radiotherapy treatment at least 6 months before study enrollement.
* Patients who are able to read, understand, and complete the questionnaire.
* Patients over 18 years of age.

Exclusion Criteria:

Acute Phase

* Patients who are unable to properly use the products.
* Patients who do not consent to participate in the study.
* Patients who were being treated for another type of cancer.

Chronic Phase

* Patients using medications such as pilocarpine, cevimeline, etc., to treat xerostomia.
* Patients who do not consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
Acute-phase 1: Frequency of severe oral mucositis (grades 3-4) in Head & Neck radiated patients (with or without concomitant chemotherapy) using a novel topical composition assessed objectively by the clinician | Six weeks during radiotherapy.
  Frequency of severe oral mucositis (grades 3-4) measured with the World Health Organization (WHO) mucositis scale, assessed at weekly intervals during 6 weeks of radiotherapy.
  Oral mucositis will be objectively assessed by clinician, based on observation of mucosa tissue damage, pain and difficulties in swallowing from grade 0 to 4, where grade 0 is the best health score and grade 4 is the worst health score. Precisely, grade 0 means no tissue injury nor pain nor difficulty in swallowing, grade 1 means presence of erythema, soreness but not difficulty in swallowing, grade 2 means presence of ulcers with or without erythema, moderate pain but able to eat solids, grade 3 means confluent ulceration with severe pain and not able to eat solids and grade 4 means deep ulcerations and/or necrotic injury, extreme pain and unable to eat solids/drink. Grades 3 and 4 are defined as severe oral mucositis (SOM).
Chronic-phase 2: Changes in long-term quality of life of radiated Head & Neck cancer patients (with or without concomitant chemotherapy) after 1 month of use of the tested composition. | One month of use of the tested product.
  Comparison of late symptoms perceived by the patient through the PROMs validated Spanish version of the University of Washington Quality of Life questionnaire (UW-QOL) before (baseline) and after 1 month using the tested composition, starting 6 months after radiotherapy completion.
  The UW-QOL questionnaire will be filled by patients at baseline and after 1 month of use of the tested composition where the possible response options (from 3 to 6) to the 12 single question domains, are scaled evenly from 0 (worst) to 100 (best) according to the hierarchy of response.

SECONDARY OUTCOMES:
Time to onset of severe oral mucositis (grades 3-4) in Head & Neck radiated patients (with or without concomitant chemotherapy) using XCM-OM118, assessed both objectively by the clinician and subjectively reported by the patient. | Six weeks during radiotherapy.
  Time to onset of severe oral mucositis (grades 3-4) determined through both objective clinical assessments and patient-reported subjective symptoms, along the 6 weeks of radiotherapy.
Comparison between physician's (objective) and patient's (subjective) perception of oral mucositis severity during treatment week by week. | Six weeks during radiotherapy.
  WHO scale will be used by clinician to objectively assess oral mucositis (OM) based on physician's observation of mucosa tissue damage, pain and difficulties in swallowing (grade 0 to grade 4) along 6 weeks of radiotherapy (RT).
  Patient reported outcomes, regarding pain and difficulties in swallowing, from grade 0 (no pain, nor difficulty in swallowing), 1 (soreness but not difficulty in swallowing), 2 (moderate pain but able to eat solids), 3 (severe pain and not able to eat solids) to grade 4 (extreme pain and unable to oral diet), will be recovered during an interview at time of visit to the unit at weekly intervals along the 6 weeks of RT.
  Evaluation of possible differences between objective and subjective OM severity data will be performed by calculating the agreement proportion and the Spearman´s rho coefficient.

OTHER OUTCOMES:
Comparison of oral mucositis severity in patients receiving radiotherapy vs patients receiving radiotherapy plus chemotherapy, with both groups using a novel topical composition | Six weeks during radiotherapy.
  Oral mucositis severity will be assessed in patients receiving radiotherapy vs patients receiving radiotherapy plus chemotherapy using both objective evaluations.
  Oral mucositis will be objectively assessed by clinician, based on observation of mucosa tissue damage, pain and difficulties in swallowing, from grade 0 (no tissue injury, no pain, nor difficulty in swallowing), grade 1 (presence of erythema, soreness but not difficulty in swallowing), grade 2 (presence of ulcers with or without erythema, moderate pain but able to eat solids), grade 3 (confluent ulceration, severe pain and not able to eat solids) to grade 4 (deep ulcerations and/or necrotic injury, extreme pain and unable to oral diet) at weekly intervals along the 6 weeks of radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Rodríguez-Vilaboa del Cura, Study Chair
Locations (1):
- Mucosa Innovations S.L., Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodriguez-Agurto A, Bravo M, Magan-Fernandez A, Lopez-Toruno A, Munoz R, Ferrer J, Mesa F. Randomized clinical trial on the clinical effects of a toothpaste containing extra virgin olive oil, xylitol, and betaine in gingivitis. Sci Rep. 2023 Apr 18;13(1):6294. doi: 10.1038/s41598-023-33521-4. PMID 37072503
- [Result] Nazar G, Garmendia ML, Royer M, McDowell JA, Weymuller EA Jr, Yueh B. Spanish validation of the University of Washington Quality of Life questionnaire for head and neck cancer patients. Otolaryngol Head Neck Surg. 2010 Dec;143(6):801-7, 807.e1-2. doi: 10.1016/j.otohns.2010.08.008. PMID 21109081
- [Result] Elting LS, Keefe DM, Sonis ST, Garden AS, Spijkervet FK, Barasch A, Tishler RB, Canty TP, Kudrimoti MK, Vera-Llonch M; Burden of Illness Head and Neck Writing Committee. Patient-reported measurements of oral mucositis in head and neck cancer patients treated with radiotherapy with or without chemotherapy: demonstration of increased frequency, severity, resistance to palliation, and impact on quality of life. Cancer. 2008 Nov 15;113(10):2704-13. doi: 10.1002/cncr.23898. PMID 18973181